CLINICAL TRIAL: NCT04105946
Title: Opioid Free Anesthesia Versus Conventional Total Intravenous Anesthesia for ENT Surgery
Brief Title: Opioid Free Anesthesia in ENT Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OFA in ENT
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Functional Endoscopic Sinus Surgery
Keywords: FESS; Opioid Free Anesthesia; Opioid Consumption
MeSH Terms: interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OFA Group (Active Comparator): patients undergoing FESS under opiod free anesthesia
  Interventions: Drug: Dexmedetomidine
- TIVA Group (Active Comparator): patients undergoing FESS under total intravenous anesthesia
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine administration intraoperatively in combination with other drugs used in OFA
  Arms: OFA Group
Drug: Remifentanil — remifentanil administration intraoperatively in combination with other drugs used in TIVA
  Arms: TIVA Group

SUMMARY:
Opioid Free Anesthesia (OFA) - which has been applied mainly in bariatric surgery - has begun to receive more and more attention and to obtain fanatical supporters versus conventional anesthesia. The advantages of this type of anesthesia are mainly achieved by the action and effect of the various drugs that compose it.

Functional Endoscopic Sinus Surgery is performed in cases where sinusitis or its complications are difficult to treat with medication. With special cameras and endoscopes, the narrow anatomical regions of the sinus can be depicted and precisely surgically approached. Usually surgery is conducted under general anesthesia. According to the literature, total intravenous anesthesia should be used for sinus surgery to achieve blood pressure control as well as controlled hypotension to prevent intraoperative bleeding. Most of the studies agree that the best type of anesthesia for this type of surgery is total intravenous anesthesia. When it comes to Opioid Free Anesthesia in FESS, there are not many studies, except of some studies that don't use solely Opioid Free Anesthesia but some of the drugs that consist it.

Patients scheduled for elective Functional Endoscopic Sinus Surgery will be randomised in two groups. One receiving OFA and one receiving TIVA.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 - 75 years old
* Elective FESS

Exclusion Criteria:

1. Patients < 18 or >75 years of age
2. Patients who can't read of speak the Greek language
3. Patients with psychiatric disorders
4. Patients with atrioventricular block in ECG
5. Patients with musculoskeletal disorders
6. Patients with coronary artery disease
7. Patients uncapable of giving informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pain management | 48 hours
  Visual Analogue Scale score for pain after FESS
Intraoperative bleeding in the surgical field | intraoperatively
  Surgeon bleeding scale 0-3 for bleeding in the operative field

SECONDARY OUTCOMES:
Patient Satisfaction | 48 hours
  Quality of recovery questionnaire for patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Elena Arnaoutoglou, MD, PhD, Study Chair — University of Thessaly; Ioannis Chatzioannou, MD, PhD, Study Director — University of Thessaly; Dimitra Papaspirou, MD, Principal Investigator — University Hospital of Larissa
Locations (1):
- Univeristy of Thessaly, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No